CLINICAL TRIAL: NCT06414291
Title: Rehydration Efficiency During Ad-libitum Fluid Intake
Acronym: LIV-D2O
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Stavros Kavouras, Professor & Assistant Dean, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: FP00039672
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Who Masked: Participant
Masking Description: non labeled bottles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Water (Placebo Comparator): Rehydration with low mineral content bottle water
  Interventions: Other: Plain Water
- Carbohydrate Electrolyte solution (Experimental): Drink with 22 grams of carbohydrate, 1020 milligrams of sodium, and 760 milligrams of potassium per liter. Hydration multiplier liquid IV
  Interventions: Other: Liquid IV Hydration Multiplier
- Low Sugar electrolyte solution (Experimental): 10 grams of carbohydrate, 1060 milligrams of sodium, and 760 milligrams of potassium per liter. Sugar free Liquid IV
  Interventions: Other: Liquid IV Sugar Free

INTERVENTIONS:
Other: Plain Water — Plain water without calories, sweetener, or electolytes
  Arms: Water
Other: Liquid IV Hydration Multiplier — Drink with 22 grams of carbohydrate, 1020 milligrams of sodium, and 760 milligrams of potassium per liter. Hydration multiplier liquid IV
  Arms: Carbohydrate Electrolyte solution
Other: Liquid IV Sugar Free — 10 grams of carbohydrate, 1060 milligrams of sodium, and 760 milligrams of potassium per liter. Sugar free Liquid IV
  Arms: Low Sugar electrolyte solution

SUMMARY:
It is well established that rehydration with a carbohydrate-electrolyte solution is more effective in comparison to plain water. This is primarily based on the sodium-glucose co transporter, based on which the world health organization has based its oral rehydration solution recommendations. Also, rehydration with a solution that includes sodium and glucose plasma osmolality should not drop as much as it happens during rehydration with water. As a result, we should have higher fluid intake due to higher thirst perception and lower urinary output due to higher levels of vasopressin.

The present study aims to examine the effectiveness of a electrolyte-glucose drink on rehydration following exercise-induced dehydration.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Training at least 2 times per week
* stable weight for the last 2 months (fluctuation less than 5 pounds)

Exclusion Criteria:

* Night shifting work
* Thyroid medication
* Bariatric surgery
* Cardiovascular disease
* Renal disease
* Hepatic disease
* Participating in another study at the same time
* Bodyweight over 110 pounds

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Total fluid intake | 4 hours of rehydration
  Total amount of fluid ingested
Net fluid balance | at 4 hours of the rehydration period
  amount of water retained during the rehydration period
Net fluid balance | at 3 hours of the rehydration period
  amount of water retained during the rehydration period
Rate of absorption | during the first 30 minutes of rehydration
  The rate of Deuterium appearance in the blood during 30 minutes of rehydration
Rate of absorption | during the first 60 minutes of rehydration
  The rate of Deuterium appearance in the blood during 60 minutes of rehydration
Rate of absorption | during the first 120 minutes of rehydration
  The rate of Deuterium appearance in the blood during 120 minutes of rehydration
Rate of absorption | during the first 180 minutes of rehydration
  The rate of Deuterium appearance in the blood during 180 minutes of rehydration
Rate of absorption | during the first 240 minutes of rehydration
  The rate of Deuterium appearance in the blood during 240 minutes of rehydration
Cumulative urine output | during the first 3 hours of rehydration
  Total amount of urine output during rehydration
Cumulative urine output | during the first 4 hours of rehydration
  Total amount of urine output during rehydration

SECONDARY OUTCOMES:
Plasma copeptin | at 30 minutes, 1 hour, 2 hours, 3 hours and 4 hours of the rehydration period
  Plasam Copeptin during rehydration
Plasma volume | at 30 minutes, 1 hour, 2 hours, 3 hours and 4 hours of the rehydration period
  percent of plasma volume recovery during the rehydration
Free water Clearance | at 30 minutes, 1 hour, 2 hours, 3 hours and 4 hours of the rehydration period
  Free water clearance calculated based on plasma and urine osmolality
Free Osmotic Clearance | at 30 minutes, 1 hour, 2 hours, 3 hours and 4 hours of the rehydration period
  Free Osmotic clearance calculated based on plasma and urine osmolality
Thirst | at 30 minutes, 1 hour, 2 hours, 3 hours and 4 hours of the rehydration period
  Thirst estimated with a visual analog scale from 0-125 millimeters with higher value indicating greater perception
Stomach fullness | at 30 minutes, 1 hour, 2 hours, 3 hours and 4 hours of the rehydration period
  Stomach fullness estimated with a visual analog scale from 0-125 millimeters with higher value indicating greater perception
Taste Likeness | at 30 minutes, 1 hour, 2 hours, 3 hours and 4 hours of the rehydration period
  Taste Likeness estimated with a visual analog scale from 0-125 millimeters with higher value indicating greater perception

CONTACTS AND LOCATIONS:
Locations (1):
- Interdisciplinary Science and Technology Building 8, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No